CLINICAL TRIAL: NCT04927923
Title: The Effect of Hope-Focused Motivational Interview on Depression, Anxiety, Stress and Hope Levels of Individuals Receiving Hemodialysis Treatment
Brief Title: The Effect of Hope-focused Motivational Interview on Individuals Receiving Hemodialysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serife Bilge Duran (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor-Investigator, Serife Bilge Duran, Principal Investigator, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5580
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Motivation; Hope; Stress; Anxiety; Depression
Keywords: HOPE; PSYCIATRIC NURSING; Motivational Interview
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled, pretest-posttest control group
Who Masked: Participant
Masking Description: Pre-test will be applied to all individuals determined according to the inclusion and exclusion criteria. After the pre-test application, the envelope method will be used to determine the individuals who will form the experimental and control groups. 1 for the experimental group in 22 envelopes and 2 for the control group in the other 22 envelopes and all of them will be stored in a box. After each patient pulls the envelope, their group will be determined and the envelope will not be thrown back into the box. The researcher who will apply the intervention and evaluate the data in this planned study is the same person. It will be ensured that only the individuals involved in the research do not learn the group they are in, and one-way blinding will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hope-focused motivational interview-experimental group (Active Comparator): * Volunteering to participate in research
  * Being over the age of 18
  * Being able to read and write
  Interventions: Other: hope-focused motivational interview
- control group (No Intervention): * Volunteering to participate in research
  * Being over the age of 18
  * Being able to read and write

INTERVENTIONS:
Other: hope-focused motivational interview — The eight-week hope-focused motivational interview will be applied to each individual individually during dialysis treatment. Within the scope of the study, a hope tree will be created for each individual together with the patients to be used in the evaluation process of the interview sessions. Through the hope tree, it is aimed for the individual to set goals, to discover the obstacles and solutions in achieving these goals.
  Arms: hope-focused motivational interview-experimental group

SUMMARY:
Chronic kidney failure (CRF) is an important health problem in the world and in our country. The use of hemodialysis as a treatment method has prolonged the life span of individuals with CRF; challenging and long treatment processes make the individual at risk for mental illnesses. It is an inevitable need to carry out psychosocial interventions to protect and improve the mental health of individuals, to ensure their adaptation to treatment processes, and to support them in coping with the difficulties they encounter. It is predicted that hope-focused motivational interviewing, which is a hope-enhancing intervention based on Snyder's Hope Theory, will be effective for individuals with low hope levels. In this study, it was aimed to evaluate the protocol suitability of the research. This study is a single blind, randomized controlled trial. The universe of the research will consist of 44 individuals coming for treatment in the Hemodialysis Unit. The study will be carried out in the Hemodialysis Clinic between September 2021 and December 2022. Within the scope of the protocol, a preliminary application was made with two individuals. Research data will be obtained by using sociodemographic data form, Depression Anxiety Stress Scale, Continuous Hope Scale. In the study, it was planned to apply hope-focused motivational interviews to the experimental group as one-hour sessions per week with face-to-face interviews for 8 weeks, while no intervention was made to the control group. Each session has goals and assignments for goals. Within the scope of the study, a hope tree will be created for everyone together with the patients to be used in the evaluation process of the interview sessions. Through the hope tree, it is aimed for the individual to set goals and discover the obstacles and solutions in reaching these goals. At the end of 8 weeks, the final test will be applied to the experimental and control groups. Following the post-test application, follow-up is planned at the end of the first month. The pre-application of the eight-week application protocol created for the purpose was made with two individuals. As a result of the preliminary application, it was observed that the stress, anxiety and depression levels of the individuals decreased and their hope levels increased. As a result of the preliminary application, it was concluded that the steps of the prepared application protocol were suitable for the study in line with the purpose determined with this patient group, and the protocol was transferred to the application phase as it was. It is thought that the results obtained from the research will contribute to the literature.

DETAILED DESCRIPTION:
Chronic kidney failure is an important health problem in the world and in our country. If crf is not diagnosed early and intervened in a timely manner, a picture called end-stage renal disease emerges and compels individuals to undergo dialysis treatment. This high-cost treatment makes individuals dependent on the health institution on certain days and hours of the week and negatively affects the quality of life of the individuals. High morbidity rates and poor quality of life also negatively affect the family and social life of these patients and hinder their economic productivity. Dialysis or kidney transplantation treatments are required for patients with esrd to survive. Since it is difficult to provide suitable conditions (donor finding, economic, etc.) For kidney transplantation, the predominant treatment method all over the world is hemodialysis with a rate of approximately 90 percent, although there are some differences between countries. The prevalence of end-stage renal disease requiring renal replacement therapy in turkey is 988.4 per million population. When looking at the type of rrt of all patients who received rrt at the end of 2018, it is seen that 74.82% received hemodialysis treatment. With the use of hemodialysis treatment as a treatment method for individuals with a diagnosis of crf, their lifespan has been prolonged, however, the type of treatment and the constant dependence on the hospital caused the psychosocial problems of individuals to increase. hemodialysis treatment patients become dependent on dialysis machines, healthcare professionals and family members throughout the treatment process, they experience role losses and domestic problems, become a risky group in terms of mental illnesses as a result of economic difficulties due to losses and an isolated life from the society. The most common mental problems in hemodialysis treatment patients; depression, restriction of social life, anxiety of losing independence, anxiety and hopelessness. Therefore, patients' adaptation to treatment processes and coping with the difficulties they encounter necessitate psychosocial interventions.

According to Babur, Abram grouped the reactions of individuals who received hemodialysis treatment treatment into five periods. He named the first period as "Uremic Period". In this period, the individual has not started dialysis yet, and with the diagnosis of CRF, hopelessness, fear of death, weakness, etc. findings indicate that it can be seen. He defined the second period as the "Anxiety Period" (Beginning of Dialysis). The anxiety period is the period in which individuals experience concerns about treatment. The third period was defined as the "Honeymoon Period" (the first three weeks in dialysis), and it was emphasized that the individual feels better, apathy decreases and euphoria may be experienced with the regression of symptoms in this period. The next period is the "Depression Period". It starts with the individual realizing the situation after 8-9 dialysis. This period, in which treatment compliance difficulties and depression are common, usually lasts 3-12 months. The last period has been defined as the "Adaptation Period". During this period, the individual has gotten used to the dialysis machine and tries to return to his normal life. There are forward plans and expectations. When the characteristics of these five periods are evaluated, although each period contains its own specific emotional and behavioral responses, it is a situation that should be evaluated to develop / strengthen hope and hope. Snyder evaluated hope in two dimensions: emotional and cognitive. The first dimension, "agency", is the desire to reach the goal and the feeling of strength to achieve the goal. It includes being able to make successful decisions in achieving the past, present and future goal. The second dimension of hope is called "pathway". Pathway dimension includes the individual's belief that he or she can plan successfully to achieve his goals. Both dimensions are related to each other and increase each other's effects in a positive way. It is a healing force that promotes well-being necessary for healthy coping. Snyder stated that as a result of studies conducted with different ethnic groups, hopeful thinking is not inherited, it is learned from childhood. Therefore, he argued that hopeful thinking can be taught and enhanced. Hope has been accepted as a basic personality trait and has been defined as a fundamental resource in human life. In other words, individuals with a high level of hope have goals they want to achieve, and individuals strive to achieve these goals. The high level of hope is important in increasing the life satisfaction of individuals.

It is seen as an effective coping mechanism that makes the individual feel safe and relate to reality, increases motivation, prevents feelings of pessimism or helplessness in case of illness, and contributes to compliance with treatment. As they increase, their compliance with treatment increases and as a result, it can be effective in reducing the symptoms of the disease.

Snyder defines it as the ability to produce ways to achieve desired goals and the motivation to use these paths. They believe that if an individual has a high level of hope, they can find many ways to achieve their goals. This belief motivates the individual that good events will happen in the future. In this direction, motivational interview enables the individual to understand their problems and put them into action for change. With motivational interview, it will be easier for the individual to notice the obstacles that may occur in achieving his goal, and he will be able to make expressions that will motivate himself about his anxiety, desire, desire for change and skill. In this context, it is predicted that with a hope-oriented motivational interview, individuals will be able to recognize their goals more easily and determine their paths. Studies involving hope-enhancing intervention are based on Snyder's Hope Theory in positive psychology. Diabetes, hypertension, depression, CRF, unstable angina, In addition to individuals with chronic diseases, hope-enhancing interventions were applied to individuals with caregiver roles such as caregivers of patients diagnosed with post-traumatic stress disorder, and mothers of children diagnosed with cancer. At the same time, different segments of society, pregnant women, married students, etc. In order to examine the effects of healthy individuals on mental health. As a result of the practices that strengthen hope, depression, anxiety, and stress levels decreased in individuals, and their well-being was observed to increase. The concept of hope is also an important concept in terms of psychiatric nursing care and practices. Moore expresses hope as the heart of Psychiatric Nursing practices. Hope, which is accepted as a fundamental element of human existence, is important in terms of preventive mental health in psychiatric nursing care and practices. Therefore, increasing patients' hope has been accepted as an important intervention in medicine, nursing and mental health. In the Classification of Nursing Interventions (NIC), this intervention was included as the title of "instilling hope", and many interventions to increase and develop the hope of the individual within the scope of the intervention (Bulechek et al. Although there are descriptive studies aimed at evaluating hope in the studies conducted in the field of nursing, intervention studies specifically aimed at increasing and developing hope are limited. When the content of the limited number of studies was examined, it was seen that the effectiveness of nursing interventions in different patient groups was evaluated. Considering the psychosocial difficulties of individuals with CRF, which is a chronic disease, it is thought that conducting an intervention study with this patient group would be effective. When psychiatric nursing practices and consultation-liaison psychiatric nursing roles are evaluated within the scope of their roles, it is predicted that hope-oriented motivational interviewing can be effective in bringing and maintaining healthy life behaviors aimed at re-evaluating the lives of individuals, protecting and improving their mental health. In this context, it was aimed to determine the effect of hope-oriented motivational interview on the depression, anxiety, stress and hope levels of individuals receiving hemodialysis treatment within the scope of the study. It is thought that the results to be obtained from the research will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Being over the age of 18
* Being able to read and write

Exclusion Criteria:

* Not attending the interview for more than 2 weeks,
* Development of a medical condition that prevents interviews,
* Exercising the participant's right to withdraw from the trial at his / her own request.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Sociodemographic data form | immediately before the first interview
  In this section, besides data such as age, gender, and educational status of the individuals, there are questions regarding the findings regarding the treatment process.
Depression Anxiety Stress Scale (DASS 21) | immediately before the first interview
  The scale, which is a 4-point Likert type, consists of 7 questions each measuring "depression, stress and anxiety dimensions".
  consists of. An individual's depression sub-dimension 5 points or more, anxiety 4 points and above, stress A score of 8 or more indicates that it has a related problem.
Dispositional Hope Scale | immediately before the first interview
  The scale, which is Likert type, consists of 12 items. It has 2 sub-dimensions, Alternative Ways Thinking and Acting Thinking, and there are 4 items for each sub-dimension. One of these items is for the past, two for the present and one for the future.The score obtained from the scale is an indicator of the hope level of the individual.
  An increase in scores is interpreted as an increase in the level of hope.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS 21) | immediately after the last interview
  The scale, which is a 4-point Likert type, consists of 7 questions each measuring "depression, stress and anxiety dimensions".
  consists of. An individual's depression sub-dimension 5 points or more, anxiety 4 points and above, stress A score of 8 or more indicates that it has a related problem.
Dispositional Hope Scale | immediately after the last interview
  The scale, which is Likert type, consists of 12 items. It has 2 sub-dimensions, Alternative Ways Thinking and Acting Thinking, and there are 4 items for each sub-dimension. One of these items is for the past, two for the present and one for the future.The score obtained from the scale is an indicator of the hope level of the individual.
  An increase in scores is interpreted as an increase in the level of hope.

CONTACTS AND LOCATIONS:
Overall Officials: İLKAY KESER, Study Chair — i.keser@akdeniz.edu.tr
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the research was completed, it was deemed appropriate to share.

REFERENCES:
- [Background] Samavi SA, Najarpourian S, Javdan M. The Effectiveness of Group Hope Therapy in Labor Pain and Mental Health of Pregnant Women. Psychol Rep. 2019 Dec;122(6):2063-2073. doi: 10.1177/0033294118798625. Epub 2018 Sep 11. No abstract available. PMID 30205789
- [Background] Rahimipour M, Shahgholian N, Yazdani M. Effect of hope therapy on depression, anxiety, and stress among the patients undergoing hemodialysis. Iran J Nurs Midwifery Res. 2015 Nov-Dec;20(6):694-9. doi: 10.4103/1735-9066.170007. PMID 26793255